CLINICAL TRIAL: NCT00317746
Title: A Randomized, Placebo Controlled Trial of Citalopram for the Prevention of Depression and Its Consequences in HIV-Hepatitis C Co-infected Individuals Initiating Pegylated Interferon/Ribavirin Therapy
Brief Title: Trial of Citalopram for the Prevention of Depression
Acronym: PICCO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marina Klein (Other)
Collaborators: Ontario HIV Treatment Network (Network); Schering-Plough (Industry); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor-Investigator, Marina Klein, Study Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTN194; Schering #2229
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Depression; HIV Infections; Hepatitis C
Keywords: HIV/HCV Co-infection; Depression; Citalopram
MeSH Terms: conditions — Depression; HIV Infections; Hepatitis C | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo + PEG-interferon-alfa2b + ribavirin
  Interventions: Drug: Placebos
- Citalopram (Experimental): Citalopram + PEG-interferon-alpha2b + ribavirin
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Citalopram
  Arms: Citalopram
Drug: Placebos
  Arms: Placebo

SUMMARY:
With the improved prognosis of human immunodeficiency virus (HIV) infection, end stage liver disease due to hepatitis C (HCV) now represents a major cause of morbidity and mortality in people with HIV. Treatment for HCV has become increasingly important as a means of preventing the consequences of chronic HCV infection. Paradoxically, co-infected patients have low rates of treatment initiation and completion in large part because they have a high risk of developing neuropsychiatric symptoms while receiving PEG-interferon (PEG-IFN). There are a large number of co-infected individuals in Canada who could benefit from HCV therapy if tolerability could be improved. This trial will address whether prophylactic use of antidepressants in HIV-HCV infected patients initiating HCV therapy can prevent the development of neuropsychiatric side effects and thus permit more patients to receive full treatment for HCV.

DETAILED DESCRIPTION:
Trial design:

This study is a Canadian multicentre randomized, double-blind placebo controlled trial. We will evaluate whether prophylactic citalopram compared to symptomatic treatment of depression can significantly increase the amount of HCV therapy received in co-infected patients during the first 24 weeks. Post study follow-up will extend until 6 months after cessation of HCV therapy (up to 72 weeks) to capture information on SVR (sustained virologic response) for HCV. 76 patients will be randomized in a 1:1 ratio to citalopram or placebo. Patients will be stratified by study centre and HCV genotype. Citalopram (or placebo) will begin 3 weeks before HCV treatment at an initial dose of 10 mg per day then be increased to 20 mg per day after one week and continued throughout treatment with PEG-IFN/ribavirin (up to 48 weeks) and then tapered to discontinuation at completion of HCV therapy. The management of depression emerging in study participants is mandated in the protocol to ensure that the original treatment assignments remain blinded while allowing for all subjects to remain in the study and mimics what would take place in clinical practice.

Analysis:

The analyses will follow the intention-to-treat approach. Random regression modelling will be employed to analyse longitudinal data on adherence to prescribed PEG-IFN and ribavirin dosage at weeks 12 and 24. Survival analyses will be used to compare the two treatment groups with respect to the time to the development of depressions.

Implications:

Prophylactic antidepressants may not only prevent overt depression but may also diminish the development of sub-clinical depressed mood. Effective prevention of a broad range of neuropsychiatric symptoms by use of citalopram has the potential to diminish morbidity associated with PEG-IFN treatment and consequently allow a greater number of patients to complete full therapy. In addition, such an approach may help patients remain adherent to their HIV therapy during the course of HCV treatment which could have long-term personal and public health implications by preventing the emergence of HIV resistance. Furthermore, if shown to be an effective strategy for preventing neuropsychiatric symptoms, treatment for HCV may become more accessible to the large number of patients who may not have ready access to the frequent and intensive psychiatric monitoring, necessary for the early detection and treatment of depression that manifests on PEG-IFN.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ adults with chronic HCV infection requiring therapy and with no contraindications to PEG-IFN/ribavirin will be enrolled.

Exclusion Criteria:

* Subjects with prior suicide attempt, active depression, treatment with antidepressants within 6 months of study entry or with other psychiatric disorders will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the average proportion of PEG-IFN and ribavirin doses received in participants receiving citalopram compared with placebo | week 24
A second major objective is to compare arms with respect to the rate of moderate-to-severe depressive symptoms during the first 24 weeks of therapy. | week 12 and week 24

SECONDARY OUTCOMES:
Secondary measures will assess impact of citalopram versus placebo on anxiety, neurocognitive function, quality of life and adherence to therapy. HCV and HIV control will also be examined. | 24 weeks
Substudies aimed at understanding the pathogenesis of neuropsychiatric side effects and neurocognitive function in this population will be performed. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marina B Klein, MD, Principal Investigator — Immunodeficiency Service Montreal Chest Institute
Locations (1):
- Immunodeficiency Service Montreal Chest Institute McGill University Health Centre, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Klein MB, Lee T, Brouillette MJ, Sheehan NL, Walmsley S, Wong DK, Conway B, Hull M, Cooper C, Haidar S, Vezina S, Annable L, Young S, Zubyk W, Singer J. Citalopram for the prevention of depression and its consequences in HIV-hepatitis C coinfected individuals initiating pegylated interferon/ribavirin therapy: a multicenter randomized double-blind placebo-controlled trial. HIV Clin Trials. 2014 Jul-Aug;15(4):161-75. doi: 10.1310/hct1504-161. PMID 25143025